CLINICAL TRIAL: NCT02371083
Title: Timing of Pessary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Katie Propst, MD, Fellow, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2014-0112
Record Dates: First submitted 2015-01-16; First posted 2015-02-25 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse managed by vaginal pessary
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine (No Intervention): Subjects will continue with regular pessary care every 12 weeks.
- Extended (Experimental): Subjects will have extended time between pessary care visits which will occur every 24 weeks.
  Interventions: Other: Extended timing of pessary care

INTERVENTIONS:
Other: Extended timing of pessary care
  Arms: Extended

SUMMARY:
This is a prospective trial to investigate optimal timing of care for vaginal pessaries. A vaginal pessary is a silicone device that is placed in the vagina to support the pelvic organs of a woman who has pelvic organ prolapse. Some women are willing and able to remove their own pessary on a regular basis. In women who are either unwilling or unable to remove their own pessary, complete pessary care is provided in the urogynecology office. Complete pessary care involves regular removal and cleaning of the pessary with a vaginal examination. In our practice, the investigators typically remove vaginal pessaries and examine the vagina every 3 months in patients for whom the investigators provide complete pessary care. Interval of pessary removal varies widely between practitioners. In the literature, removal intervals vary from weekly to yearly. In this study, the investigators will randomize participants to pessary care with removal every 12 weeks or every 24 weeks.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded trial of office-based pessary care. The primary outcome of this study is vaginal epithelial abnormalities, including granulation tissue and ulceration. Secondary outcomes include participant satisfaction, degree of bother due to vaginal discharge, number of unscheduled visits and progression of pelvic organ prolapse quantification score (POPQS).

At baseline (visit 1; see "Visit Schedule", below), women who have consented to participate will be randomized 1:1 to one of two groups:

1. routine group: pessary care with removal and cleaning every 12 ± 2 weeks, or
2. extended group: pessary care with removal and cleaning every 24 ± 2 weeks.

Randomization will be performed using a randomization scheme available through Excel. Each consecutive/sequential participant will be assigned to whichever group corresponds to that sequential study entry number.

For both groups, the pessary will be removed and cleaned and a vaginal examination will be performed at every visit regardless of complaints. The only difference will be frequency of visits. All pelvic examinations will be performed by the same individual.

The study will be conducted for approximately one year, with additional time for analysis and preparation of abstract(s) and manuscript(s). Subjects' participation will consist of five visits in the routine group, three visits in the extended group. Consent to study participation will be obtained at the first visit. Visit schedule is shown below:

Visit Schedule Routine Group Visit #1, initial visit (week 0), procedures: Consent to participate, Collect Demographics, Pelvic examination /pessary removal Consent to participate Visit #2, interim visit (week 12 ± 2), procedures: Interview, Pelvic examination /pessary removal Visit #3, interim visit (week 24 ± 2), procedures: Interview, Pelvic examination /pessary removal Visit #4, interim visit (week 36 ± 2), procedures: Interview, Pelvic examination /pessary removal Visit #5, final visit (week 48 ± 2), procedures: Interview, Pelvic examination /pessary removal

Extended Group Visit #1, initial visit (week 0), procedures: Consent to participate, Collect Demographics, Pelvic examination /pessary removal Consent to participate Visit #2, interim visit (week 24 ± 2), procedures: Interview, Pelvic examination /pessary removal Visit #3, final visit (week 48 ± 2), procedures: Interview, Pelvic examination /pessary removal

Participants who are approaching the upper bound of their visit window will be reminded of the need for a visit. Those who still present outside of the window for the interim visit will be scheduled their next appointment as it would have been scheduled if they had presented for the visit at the correct time. Any such cases will be noted in the analysis and a protocol deviation form will be completed and sent to IRB. Any participant who misses three visits within the scheduled window will be withdrawn from the study.

Consent to study participation will occur at visit #1, a vaginal examination will be performed to document a pelvic organ prolapse quantification score8 (POPQS) and to exclude the presence of vaginal epithelial abnormalities (granulation tissue, erosion), or fistula and to note the presence of vaginal adhesions.

Additional data will be collected at the initial visit: age, body mass index (BMI), smoking status, history of diabetes mellitus, history of surgery for incontinence or pelvic organ prolapse, history of hysterectomy, indication for pessary use, pessary size and type, duration of pessary use of the current pessary and in total if the participant has used other pessaries in the past, whether the participant has an intimate partner, use of aspirin (ASA) and dose, use of anticoagulation therapy, parity, bother from vaginal discharge, presence of vaginal bleeding, and history of vaginal epithelial abnormalities. The investigators also will document if the participant is using hormone replacement (HRT). If the participant is using HRT, the investigators will document medication, dose, route and frequency.

Participants will be followed for 48 ± 2 weeks. At interim visits, data will be assessed for updates:

Has the participant started new medications (ASA, anticoagulation, HRT)? Is the subject bothered by vaginal discharge? Is vaginal bleeding present?

At interim visits, when a pessary is removed, a vaginal examination will be performed to evaluate for the presence of vaginal epithelial abnormalities and vaginal adhesions. When abnormalities are noted, they will be described in appearance, location, number, and size. Additionally, abnormalities will be staged using the following system:

Stage Description

1. Epithelial erythemya without epithelial breaks or presence of granulation tissue ≤1cm in size.
2. Epithelial break or erosion ≤ 0.5 cm in diameter or presence of granulation tissue >1cm in size.
3. Epithelial break or erosion 1-2cm in diameter.
4. Epithelial break or erosion > 2 cm in diameter.

If there is more than one epithelial abnormality noted, each will each be assigned a stage. The highest stage abnormality will determine the overall stage of the epithelial abnormality.

If there is a change in pessary type or size, this will be documented. If the pessary is changed to a type other than ring or gellhorn, the participant will continue in the study as scheduled. If a pessary is removed and left out of the vagina, this will be documented. At the final visit, all participants will undergo a pelvic examination with pessary removal.

Data will be collected on forms designed according to study group (routine/extended) and visit number. In the case that a participant has a pessary complaint and requires evaluation in the office outside of the scheduled visits according to their group allocation, an unscheduled visit form will be used to collect data at this visit. At an unscheduled visit, the same data will be collected as is collected at a scheduled follow-up visit. Additionally, the participant's complaint/visit reason will be described.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* age greater than 17 years
* able and willing to participate
* patients who are currently wearing a ring, gellhorn, or incontinence dish pessary to treat pelvic organ prolapse and/or incontinence

Exclusion Criteria:

* male sex
* age less than 18 years
* unable/unwilling to participate
* patients who do not wear a pessary
* patients wearing a pessary that is not a ring or a gellhorn
* presence of vaginal granulation tissue
* erosions, or fistula, patients who perform pessary self-care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
vaginal epithelial abnormalities | Routine group: change from baseline in vaginal epithelial abnormalities at 12 weeks, 24 weeks, 36 weeks, 48 weeks. Extended group: change from baseline in vaginal epithelial abnormalities at 24 weeks, 48 weeks
  this will be evaluated by vaginal examination at each study visit

SECONDARY OUTCOMES:
Patient satisfaction | final study visit (48 weeks)
  this will be evaluated at the final visit by asking patients if they preferred more or less frequent pessary visits
Degree of bother due to vaginal discharge | Routine group: change from baseline in degree of bother due to vaginal discharge at 12 weeks, 24 weeks, 36 weeks, 48 weeks. Extended group: change from baseline in degree of bother due to vaginal discharge at 24 weeks, 48 weeks
  this will be assessed by asking participants how bothersome is vaginal discharge on a 5-point likert scale
Progression of Pelvic Organ Prolapse Quantification Score | Change from baseline in pelvic organ prolapse quantification score at final study visit (48 weeks)
  this will be evaluated by measuring a pelvic organ prolapse quantification score on physical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Urogynecology Division, Hartford, Connecticut, United States

REFERENCES:
- [Derived] Bugge C, Adams EJ, Gopinath D, Stewart F, Dembinsky M, Sobiesuo P, Kearney R. Pessaries (mechanical devices) for managing pelvic organ prolapse in women. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD004010. doi: 10.1002/14651858.CD004010.pub4. PMID 33207004
- [Derived] Propst K, Mellen C, O'Sullivan DM, Tulikangas PK. Timing of Office-Based Pessary Care: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jan;135(1):100-105. doi: 10.1097/AOG.0000000000003580. PMID 31809432